CLINICAL TRIAL: NCT05538299
Title: Silicosis Prevalence and Related Knowledge, Attitudes and Practices Among Mine Workers in Rural Rwanda
Brief Title: Silicosis Treatment, Action, Screening and Surveillance in Rwanda Trials
Acronym: STARSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samuel Hatfield (Other)
Responsible Party: Sponsor-Investigator, Samuel Hatfield, Co-Investigator, Partners in Health
Organization: Partners in Health (Other)
Other Study IDs: IMB-sil1
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Silicosis; Silicotic Fibrosis (Massive) of Lung
MeSH Terms: conditions — Silicosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaire, KAP — Diagnostic studies including questionaire, CXR, spirometry, clinical assesment, occupational safety training
  Other Names: diagnostic

SUMMARY:
Silicosis is the most prevalent occupational lung disease in low- and middle-income countries (LMICs) with "tens of millions" estimated to suffer from the disease according to the World Health Organization (WHO). To date, there is little published data on silicosis in LMICs and the burden of silicosis in Rwanda has not been well-defined. Silicosis among local mine workers is a common reason for hospitalization and death at Rwinkwavu District Hospital, located in Rwanda's Kayonza District.

The objectives of this study are:

1. To assess the prevalence of silicosis among workers in four mines located in the Kayonza District of Rwanda
2. To adapt a validated screening tool testing in Dutch construction workers for Rwandan miners
3. To implement an occupational health education program and assess the change of before and after intervention that target towards proper use of PPE and individual risk assessment in mine workers using knowledge-attitudes-practice tool

DETAILED DESCRIPTION:
Based on the clinical experience of the investigators and their network, silicosis morbidity and mortality have been consistently encountered among Rwandans with dust and mining exposure, however Rwanda currently lacks an existing body of data on current silicosis prevalence and a surveillance system for ongoing monitoring and interventions. According to the WHO, disease surveillance programs should include periodic identification and collection of health information, evaluation and interpretation of the information, and reporting and interventions for the purpose of prevention. The goal of surveillance is to monitor the trends in disease incidence over time across a particular domain, define the magnitude or relative magnitude of a problem and target and evaluate interventions. Here, the investigators propose a study of silicosis-related data from mine workers in Rwanda's Eastern Province through the development of a silicosis surveillance and health education program at Rwinkwavu District Hospital.

Methodology:

Study setting:

This study will be conducted in four sectors (Rwinkwavu, Murama, Ruramira, and Mwiri) of Kayonza district in eastern Rwanda. There are 9 [Migera, Gihinga, Nyarunazi, Gahengeli, Gashushyi, Rutonde, Raveri, Bugambira, Rukira] mining sites in Rwinkwavu, Murama, Ruramira and Mwiri, and all mining activities in these sites are supervised by Wolfram Mining and Processing LTD. All these sectors are located in the Rwinkwavu District Hospital catchment area.

Study design:

This will be a combination of a cross-sectional study to determine the prevalence of silicosis and a pre- and post-design to assess the silicosis-related knowledge, attitudes and practices (KAP) among mining workers before and after the implementation of a health education program.

The study design will be cross-sectional study. There are three main objectives: silicosis prevalence; baseline silicosis-related knowledge, attitudes and practices (KAP); and the impact of occupational health education. A team of clinical and public health professionals affiliated with Partners In Health/Inshuti Mu Buzima and Rwinkwavu District Hospital will carry out the study with data collection assistance. The preparation phase will involve contacting and establishing agreements with stakeholders from key organizations including Rwinkwavu District Hospital, Wolfram Mining and Processing Ltd., University of Rwanda and Partners in Health/Inshuti Mu Buzima. This phase will involve training data collectors and recruiting study subjects. The study execution phase will firstly consist of a cross-sectional analysis of silicosis prevalence, adapting a validated silicosis questionnaire screening tool to the target study population and performing spirometry and chest radiography to all targeted miners [Suarthana, Eva, et al. "A Simple Diagnostic Model for Ruling Out Pneumoconiosis among Construction Workers." Occupational and Environmental Medicine, JSTOR]. This screening tool for ruling out occupational pneumoconiosis, and silicosis specifically, was developed by researchers in the Netherlands. The investigators will adapt and validate the use of this screening tool to Rwandan mine workers by comparing the screening results with objective spirometry and chest radiograph findings on all subjects who have spent at least one cumulative year working directly with mining products. Secondly, the execution phase will involve an analysis of existing silicosis related KAP and the delivery of targeted occupational health education to study subjects followed by a reassessment of knowledge and attitudes. The Investigators will perform initial education program and KAP survey at the time of questionnaire-based screening with re-assessment at 2-week time point. There are approximately 995 mine workers in the catchment area of this study and the investigators' goal is to try and involve all of these stakeholders. Baseline KAP survey will be done prior to this health education program on PPE, environmental controls and personal safety assessment and deployment of the screening questionnaire. Silicosis related KAP data will be collected by skilled data collectors after a two-week training program.

Study population:

All eligible mine workers in Kayonza District in four sectors including: Rwinkwavu, Murama, Ruramira, and Mwiri sectors, located in the Rwinkwavu DH catchment area will be included in the study. Those miners with potential risk for RCS exposure, including those who handle mining either underground or above ground will be included. People who work in WOLFRAM administration (office) and never directly touch mines will not be included.

Study sample:

For the aim to determine the prevalence of silicosis, The investigators used the single population proportion formula to calculate the required sample size. With the existing literature that silicosis prevalence among high-risk populations in LMICs may range between 30-50% [Trapido, A.S. et al (1998) Prevalence of occupational lung disease in a random sample of former mineworkers, Libode District, Eastern Cape Province, South Africa. American Journal of Industrial Medicine, Antão VC, Pinheiro GA, et al., High prevalence of silicosis among stone carvers in Brazil. Am J Ind Med. 2004], The investigators used the most conservative estimate of 50% for a maximum sample size, with a level of confidence of 95%, 0.8 power and a level of precision of +/- 10% - a sample of 189 individuals will be required. For the silicosis-related KAP part of this study, the investigators also used the most conservative estimate of 50%, a 95% confidence level, and a 0.8 power to detect a 20% difference from pre- to post-intervention. This gave us a required total sample size of 186 individuals (a minimum sample of 93 individuals will be required for the pre- and post-survey), however the required sample size would increase to 224 individuals (112 individuals in each survey) after accounting for a 20% non-response rate. The investigators estimate the study sample to be around 995 mine workers, so there will be ample participants to conduct this study.

The investigators' goal is to sample the complete mining population so as to obtain accurate prevalence of the full cohort of miners within the RDH catchment area, which may also allow us to detect asymptomatic disease in certain miners, and to enroll these patients in future surveillance programs. Additionally, validation of a screening questionnaire in Rwanda will allow us to deploy a low-cost tool in the rural health network to identify additional early cases of silicosis in the community

ELIGIBILITY:
Inclusion Criteria:

* Miners with greater than 1 year of potential exposure to respirable crystalline silica within the defined catchment area of the study

Exclusion Criteria:

* non-mining (administrative, low risk of exposure) workers within the WOLFRAM (mining company) catchment area

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible mine workers in Kayonza District in four sectors including: Rwinkwavu, Murama, Ruramira, and Mwiri sectors, located in the Rwinkwavu DH catchment area will be included in the study. Those miners with potential risk for RCS exposure, including those who handle mining either underground or above ground will be included. People who work in WOLFRAM administration (office) and never directly touch mines will not be included.
Sampling Method: Probability Sample
Enrollment: 995 (Estimated)
Dates: Start 2022-07-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Silicosis Prevalence | 6 months
  Estimate Silicosis prevalence in the Eastern Province of Rwanda

SECONDARY OUTCOMES:
Questionnaire Validation | 1 year
  Validate Questionnaire originated in Europe for use in occupational health screening in Rwanda
Knowledge, Action, Prevelence | 1 year
  Obtain data on knowledge, action and practice for individual, administrative and engineering controls for spread of silica dust in mines in Eastern Rwanda

CONTACTS AND LOCATIONS:
Overall Officials: Innocent Kamali, Principal Investigator — Partners in Health
Locations (1):
- Rwinkwavu District Hospital, Rwinkwavu, Kayonza, Rwanda

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared publicly for further research involving silicosis 6-9 months following the completion of this trial
Supporting Information: Study Protocol, SAP, CSR
Time Frame: the investigators plan to make data public 6-9 months following the completion of the study and accessible for up to 3 years
Access Criteria: Access will be granted to qualified and interested researchers who approach the investigators directly following the conclusion of the study. Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). Data will be de-identified for protection of PHI

REFERENCES:
- [Background] Suarthana E, Moons KG, Heederik D, Meijer E. A simple diagnostic model for ruling out pneumoconiosis among construction workers. Occup Environ Med. 2007 Sep;64(9):595-601. doi: 10.1136/oem.2006.027904. Epub 2007 Apr 4. PMID 17409183

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05538299/Prot_SAP_001.pdf